CLINICAL TRIAL: NCT01741038
Title: A Phase II/III, Randomized, Open Label, Controlled, Two Arm Study Comparing Overall Survival of AlloStim® Combined With Cryoablation to a Physician's Choice Combined With Cryoablation in 3rd Line Treatment for Metastatic Colorectal Cancer
Brief Title: AlloStim® In-Situ Vaccine in Pre-Treated Metastatic Colorectal Cancer
Status: Withdrawn | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: moved study to USA
Sponsor: Mirror Biologics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ITL-008-INSTAVAC-CRC
Record Dates: First submitted 2012-11-29; First posted 2012-12-04 (Estimated); Last update posted 2020-01-22 (Actual); Status verified 2016-08

CONDITIONS: Metastatic Colorectal Cancer
Keywords: Cancer Vaccine; AlloStim®; Immunovative; Immunotherapy; Allogeneic Cell Therapy; Cryoablation
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Cryosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- AlloStim® treatment (Experimental): The treatment schedule includes: (1) the priming step with two ID AlloStim® injections (Days 0 and 3), an additional two ID injections followed by IV infusion of AlloStim® (Days 7 and 10); (2) the vaccination step with cryoablation of a single metastatic lesion followed by injection of AlloStim® into the ablated tumor and IV infusion of AlloStim® on protocol day 14, followed by IV infusion of AlloStim® on Day 17 (3) the activation step with an IV study drug infusion on Day 21 and (4) the booster step with IV booster infusions of AlloStim® on days 49 and 77. Additional booster infusions can be administered monthly at the discretion of the Investigator.
  Interventions: Biological: AlloStim®; Procedure: cryoablation
- Physician's Choice (PC) (Other): All subjects will be assigned Physician's Choice (PC) therapy. PC can consist of best supportive care (BSC) or any US-FDA-approved cancer drug (e.g. Cetuximab) administrated as a monotherapy at the manufacturer's recommended dose. The treatment schedule shall be prospectively determined and administered as tolerated.
  Interventions: Procedure: cryoablation; Other: Physician's Choice (PC)

INTERVENTIONS:
Biological: AlloStim® — AlloStim® is derived from the blood of normal blood donors and is intentionally mismatched to the recipient. CD4+ T-cells are separated from the blood and differentiated and expanded for 9-days in culture to make an intermediary called T-Stim. AlloStim is made by incubating T-Stim cells for 4h with antibody coated microbeads. The cells with the beads still attached are suspended in infusion media and loaded into syringes. The syringes are shipped refrigerated to the point-of-care.
  Arms: AlloStim® treatment
Procedure: cryoablation — percutaneous ablation of a single metastatic tumor lesion usually in liver. The procedure is conducted under CT or ultrasound image-guidance.
Other: Physician's Choice (PC) — Physician's Choice therapy can consist of best supportive care (BSC) or any US-FDA approved cancer drug (e.g. Cetuximab) administrated as a monotherapy at the manufacturer's recommended dose. The treatment schedule shall be prospectively determined and administered as tolerated
  Other Names: best supportive care; monotherapy (e.g.Cetuximab)
  Arms: Physician's Choice (PC)

SUMMARY:
This is a personalized anti-cancer vaccine protocol which includes an in-situ (in the body) cancer vaccine step which combines killing a single metastatic tumor lesion by use of cryoablation in order to cause the release of tumor-specific markers to the immune system and then injecting bioengineered allogeneic immune cells (AlloStim) into the lesion as an adjuvant in order to modulate the immune response and educate the immune system to kill other tumor cells where ever they reside in the body.

DETAILED DESCRIPTION:
Colorectal cancer (CRC) ranks as the third most common cancer worldwide. Metastasis is the main reason of death in CRC patients. The current drugs used to treat colorectal cancer provide important treatment options for patients, their limitations including drug resistance, poor efficacy and severe side effects. Development of new therapeutic strategies for KRAS mutant as well as BRAF mutant tumors are therefore highly needed in order to offer a new category of drug (immunotherapy). This study targets the population of mCRC patients that have progressed after two lines of chemotherapy and are not eligible for targeted therapies due to a mutation in KRAS or BRAF.

This is a Phase II/III, randomized, open-label, multicenter, controlled, two arm study designed to determine the efficacy in terms of OS and the safety of the InSituVax (AlloStim+ Cryoablation) personalized in-situ anti-cancer vaccine protocol (Treatment Arm) compared with Physician's Choice (PC) of Treatment + Cryoablation (Control Arm) in Metastatic Colorectal Cancer. Subjects are randomized 2:1 into the treatment or control arms.

ELIGIBILITY:
Inclusion Criteria:

1. Adult males and female subjects aged 18 years or older at screening visit
2. Pathological diagnosis of colorectal adenocarcinoma
3. Metastatic disease with at least one lesion in liver

   * Primary can be intact or resected
   * Metastatic lesion(s) in liver non-resectable
   * Extrahepatic disease acceptable
4. KRAS/BRAF mutant disease or KRAS wild type w/previous anti-EGFR treatment
5. At least one liver lesion able to be visualized by ultrasound and determined to be safely assessable for percutaneous cryoablation
6. Previous treatment failure of at 2 previous lines of active systemic chemotherapy for metastatic disease:

   * Previous chemotherapy must have included one line with oxaliplatin (e.g. FOLFOX) and a previous second line with irinotecan (e.g. FOLFIRI) with or without bevacizumab
   * If KRAS wild type, at least one anti-EGFR therapy in first or second line
   * Treatment failure can be due to disease progression or toxicity
   * Disease progression on 2nd line therapy must be documented radiologically and have occurred during or within 30 days following the last administration of 2nd line chemotherapy
7. ECOG performance score: 0-1
8. Adequate hematological function: Absolute granulocyte count ≥ 1,200/mm3, Platelet count ≥ 100,000/mm3, PT/INR ≤ 1.5 or correctable to <1.5 at time of interventional procedures, Hemoglobin ≥ 9 g/dL (may be corrected by transfusion)
9. Adequate Organ Function: Creatinine ≤ 1.5 mg/dL, Total bilirubin ≤ 1.5 times ULN, Alkaline phosphatase ≤ 2.5 times ULN, AST or SGOT ≤ 2.5 times ULN, ALT or SGPT≤2.5 times ULN
10. EKG without clinically relevant abnormalities
11. Female subjects: Not pregnant or lactating
12. Subjects with child bearing potential must agree to use adequate contraception
13. Study specific informed consent in the native language of the subject

Exclusion Criteria:

1. Peritoneal carcinomatosis
2. Moderate or severe ascites requiring medical intervention
3. Prior hepatectomy, ablation or chemoembolization of liver lesion
4. Prior pelvic radiotherapy
5. Clinical or radiological evidence of brain metastasis/leptomeningeal involvement
6. Symptomatic asthma or COPD or any lung condition requiring treatment with steroids
7. Pulmonary lymphangitis or symptomatic pleural effusion (grade ≥ 2) that results in pulmonary dysfunction requiring active treatment or oxygen saturation <92% on room air
8. Bevacizumab (Avastin®) treatment within 6 weeks of scheduled cryoablation
9. No Regorafenib prior to or during the Study Period
10. Anticoagulant medication for concomitant medical condition (unless can be safely discontinued for invasive cryoablation, biopsy and intratumoral injection procedures)
11. Prior allogeneic bone marrow/stem cell or solid organ transplant
12. Chronic use (>2 weeks) of greater than physiologic doses of a corticosteroid agent (dose equivalent to>5 mg/day of prednisone) within 30 days of the 1st day of study treatment

    o Topical corticosteroids are permitted
13. Prior diagnosis of an active autoimmune disease (e.g., rheumatoid arthritis, multiple sclerosis, autoimmune thyroid disease, uveitis). Well controlled Type I diabetes allowed.
14. Prior experimental therapy
15. History of blood transfusion reactions
16. Known allergy to bovine products
17. Progressive viral or bacterial infection

    o All infections must be resolved and the patient must remain afebrile for seven days without antibiotics prior to being placed on study
18. Cardiac disease of symptomatic nature
19. History of HIV positivity or AIDS
20. Concurrent medication known to interfere with platelet function or coagulation (e.g., aspirin, ibuprofen, clopidogrel, or warfarin) unless such medications can be discontinued for an appropriate time period based on the drug half-life and known activity (e.g., aspirin for 7 days) prior to cryoablation procedure
21. History of severe hypersensitivity to monoclonal antibody drugs or any contraindication to any of the study drugs
22. Psychiatric or addictive disorders or other condition that, in the opinion of the investigator, would preclude study participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-12 (Estimated); Primary Completion 2019-12 (Estimated); Study Completion 2020-10 (Estimated)

PRIMARY OUTCOMES:
Overall Survival | from randomization within 30 days of accrual to death for any cause followed for up to 2 years from date of randomization
  To assess whether cryoablation combined with AlloStim treatment (arm 1) provides an overall survival (OS) advantage when compared to treatment with cryoablation combined with physician's choice (arm 2).

SECONDARY OUTCOMES:
Safety | 168 days from randomization
  Safety will be evaluated by physical exam, changes in laboratory values and patient reported symptoms
Health-Related Quality of Life (HRQoL) | 168 days from randomization
  To assess change in HRQoL between treatment arms

OTHER OUTCOMES:
Immunological Response | 168 days from randomization
  blood samples will be evaluated for immunological response and a determination made as to whether immunological response correlates with survival
Longitudinal changes in tumor burden | 168 days from randomization
  To document the longitudinal changes in tumor burden by Response Evaluation Criteria in Solid Tumors (RECIST) and Immune-Related Response Criteria (irRC)

CONTACTS AND LOCATIONS:
Overall Officials: Wirote Lausoontornsiri, MD, Principal Investigator — National Cancer Institute of Thailand; Thu Bui, BS, Study Director — Mirror Biologics, Inc.
Locations (1):
- National Cancer Institute of Thailand, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Har-Noy M, Zeira M, Weiss L, Fingerut E, Or R, Slavin S. Allogeneic CD3/CD28 cross-linked Th1 memory cells provide potent adjuvant effects for active immunotherapy of leukemia/lymphoma. Leuk Res. 2009 Apr;33(4):525-38. doi: 10.1016/j.leukres.2008.08.017. Epub 2008 Oct 1. PMID 18834631
- [Background] Har-Noy M, Zeira M, Weiss L, Slavin S. Completely mismatched allogeneic CD3/CD28 cross-linked Th1 memory cells elicit anti-leukemia effects in unconditioned hosts without GVHD toxicity. Leuk Res. 2008 Dec;32(12):1903-13. doi: 10.1016/j.leukres.2008.05.007. Epub 2008 Jun 18. PMID 18565579
- [Background] Har-Noy M, Slavin S. The anti-tumor effect of allogeneic bone marrow/stem cell transplant without graft vs. host disease toxicity and without a matched donor requirement? Med Hypotheses. 2008;70(6):1186-92. doi: 10.1016/j.mehy.2007.10.008. Epub 2007 Dec 3. PMID 18054441